CLINICAL TRIAL: NCT00719953
Title: A Single-Center, Open-label Study to Assess the Efficacy of Cognitex in Elderly Subjects With Memory Impairment
Brief Title: Study to Assess the Efficacy of Cognitex
Acronym: Cognitex001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Enzymotec (Industry)
Responsible Party: Yael Richter. Project Manager, Enzymotec Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-08-NV-305-CTIL; 0305-08-TLV
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2008-07

CONDITIONS: Elderly; Memory Impairment
Keywords: Cognitex; subjects
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Cognitex — Treatment will consist of one capsule of Cognitex (Life Extension, USA), three times a day, with meals, delivering a total of 600 mg GPC, 100 mg PS-omega 3, 20 mg vinpocetine, 50 mg uridine-5'-monophosphate (disodium), 550 mg plant extracts (150 mg wild blueberry, 125 mg ashwagandha, 150 mg grape seed, 125 mg hops, ginger and rosemary). Duration: 15 weeks

SUMMARY:
A Single-Center, Open Label Study to Assess the Efficacy of Cognitex in Elderly Subjects with Memory Impairment

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give written informed consent.
2. Age: 90≥ years ≥60.
3. Gender: male and female.
4. Memory test performance within or below the mean established for adults in the computerized cognitive tool, with a maximum of four neuropsychological subtests scored 1.5 SD above the mean.
5. Language: Subjects must be able to read, write and speak Hebrew.
6. Ability to perform tests and interviews.

Exclusion Criteria:

1. Evidence of delirium, confusion, or other disturbances of consciousness.
2. Evidence of dementia.
3. Any Neurological disorder that could produce cognitive deterioration. Such disorders include Parkinson's disease, stroke, intracranial hemorrhage, local brain lesions including tumors and normal pressure hydrocephalus.
4. History of any infective or inflammatory brain disease including those of viral, fungal, or syphilitic etiologies.
5. Head injury immediately preceding cognitive deterioration.
6. Evidence of depression as determined by a the Geriatric Depression Scale (short version) score of 5 or more.
7. Current diagnosis or history of alcoholism or drug dependence.
8. Any medical disorder that could produce cognitive deterioration including renal, respiratory, cardiac, and hepatic disease, diabetes mellitus, endocrine, metabolic or hematological disturbances unless well controlled, and malignancy not in remission for more than two years
9. Use of anti-clotting or antiplatelet medications or supplements for less than two years.
10. History of clotting or platelet disorder unless well controlled.
11. Use of any supplement that may significantly affect cognitive functioning during the month prior to study initiation.
12. Use of any experimental medication within 1 month prior to screening or as concomitant medications.
13. History of hypersensitivity or allergy to soy or fish.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Professor, Principal Investigator — Tel-Aviv Sourasky Medical Center, Israel
Locations (1):
- Suorasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Richter Y, Herzog Y, Eyal I, Cohen T. Cognitex supplementation in elderly adults with memory complaints: an uncontrolled open label trial. J Diet Suppl. 2011 Jun;8(2):158-68. doi: 10.3109/19390211.2011.569514. PMID 22432687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements in senior citizens' homes, hospitals, and newspapers.
Period: Overall Study
Arm/Group | Cognitex
Started | 30
Completed | 26
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cognitex
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 72.97 (6.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  Israel | 30

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Cognitive Performance (Change From Baseline in Neuropsychological Computerized Test)
Description: The computerized neuropsychological assessment software consists of seven separate tasks: symbol spotting, pattern identification, pattern recall, digit-symbol substitution, digits span forward, digits span backward and delayed pattern recall. Based on the results obtained in the single tasks, eight cognitive composite scores are calculated including focused attention, sustained attention, memory recognition & recall, visuospatial learning, spatial short term memory, executive functions and mental flexibility.The total score range is from 0 to 100 points(0 is worse, 100 is best).
Time Frame: Base line and 12 weeks
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Cognitex
Number analyzed (Participants) | 26
Points on a scale
  Focused Attention | 3.46 (1.72)
  Sustained Attention | 13.19 (3.02)
  Memory - Recognition | 7.92 (2.13)
  Memory - Recall | 9.19 (2.44)
  VisuoSpatial Learning | 19.84 (3.78)
  Spatial Short Term Memory | 18.88 (4.62)
  Executive Functions | 18.61 (3.79)
  Mental Flexibility | 19.65 (3.80)

ADVERSE EVENTS:
Arm/Group | Cognitex
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitex (N=30)
Dirarrhea (Gastrointestinal disorders) | 2 (3) — Two patients were affected, only one event was defined as probably related.
Hypertension (Vascular disorders) | 3 (3) — Three patients were affected, two of them had a history of hypertension, and theirs events were defined as not related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No